CLINICAL TRIAL: NCT03618901
Title: A Randomized Crossover Trial: The Effects of Rock Steady Boxing vs. Sensory Attention Focused Exercise on Disease Progression for Those With Parkinson's Disease.
Brief Title: Rock Steady Boxing vs. Sensory Attention Focused Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Kishoree, Graduate Student, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MDRC2
Record Dates: First submitted 2018-07-18; First posted 2018-08-07 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The early start group: 12-weeks (intervention) followed by 12-weeks of no exercise.
  The delayed start group: 12-weeks (no exercise) followed by 12-weeks (intervention).
  This model will be used for both RSB and PD SAFEx.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rock Steady Boxing (Experimental): Non-contact boxing program.
  Interventions: Other: Rock Steady Boxing
- PD SAFEx (Active Comparator): Sensory attention focused exercise.
  Interventions: Other: PD SAFEx

INTERVENTIONS:
Other: Rock Steady Boxing — Boxing programs as offered by the Rock Steady Boxing institution,
  Arms: Rock Steady Boxing
Other: PD SAFEx — Progressive proprioception training.
  Arms: PD SAFEx

SUMMARY:
This study evaluates the effect on Rock Steady Boxing (RSB) and PD SAFEx on Parkinson's disease.

DETAILED DESCRIPTION:
Both interventions produce benefits to the PD population. PD SAFEx has been proven to improve the motor symptoms of PD. However, research still needs to be conducted on the PD specific benefits associated with RSB. As such it an RCT is necessary to compare the effects of both interventions.

ELIGIBILITY:
Inclusion Criteria:

* must be able to understand verbal instructions in English
* diagnosed with idiopathic PD by a neurologist

Exclusion Criteria:

* if diagnosed with a neurological condition other than PD
* if participated in an exercise program at least 2-weeks prior to the start of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Motor symptom improvements | change from baseline at 12 weeks
  Unified Parkinson Disease Rating Scale (UPDRS) conducted by a qualified movement disorders specialist. The maximum score is 108, the higher the score, the worse the symptoms.

SECONDARY OUTCOMES:
Quality of life assessments | change from baseline at 12 weeks
  Completion of Parkinson's Disease Questionnaire (PDQ-39). There are 8 sections: mobility (sub score 10), activities of daily living (sub score 6), emotional well-being (sub score 6), stigma (sub score 4), social support (sub score 3), cognition (sub score 4), communication (sub score 3) and bodily discomfort (sub score 3). The higher the score, the worse the symptoms.
Balance1 | change from baseline at 12 weeks
  Using the Biodex balance system. The postural stability test (PST) will be conducted. The results will be presented as actual score and standard deviation for both legs to determine an individuals ability to maintain balance. The lower the score the better.
Gait1 | change from baseline at 12 weeks
  For the timed-up-and-go test (TUG) participants will stand up, walk to the line on the floor, turn around and walk back to the chair and sit down.
Strength | change from baseline at 12 weeks
  Will be assessed using the Jamar hand dynamometer.
Cognitive Assessment 1 | change from baseline at 12 weeks
  Scale of Outcomes of Parkinson Disease (SCOPA-COG), will be used to assess memory and visuospatial function. There are 5 sections: memory learning, attention, executive functions, visuo-spatial functions and memory. The total score that can be achieved is 43 (the higher the score the better).
cognitive assessment 3 | change from baseline at 12 weeks
  Completion of Montreal Cognitive Assessment (MoCA). There are a total 30 points, the higher the score the better (26 and above is normal).
Balance 2 | change from baseline at 12 weeks
  Activities-specific Balance Confidence Scale (ABC). The total score that can be achieved is 16, the higher the percent the more self-confidence.
Cognitive assessment 2 | change from baseline at 12 weeks
  Mini-Mental State Examination (MMSE). The total score than can be achieved is otal score 30 (the higher the score the better).

OTHER OUTCOMES:
Balance3 | change from baseline at 12 weeks
  Balance will be measured using the mini- Balance Evaluation Systems Test (mini-best test). There are 4 sections: anticipatory, (sub score 6) reactive postural control (sub score 6), sensory orientation (sub score 6), dynamic gait (sub score 10). The total score that can be achieved is 28. The higher the score the better the balance.
Physical activity | change from baseline at 12 weeks
  Community Healthy Activities Model Program for Seniors (CHAMPS) is a questionnaire used to assess the weekly frequency and duration of the physical activities of seniors.
Gait 2 | change from baseline at 12 weeks
  For the 6-minute walking test (6MWT) participants will be asked to walk as far as possible for 6 minutes. The further (more laps) they are able to walk the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Research and Rehabilitation Centre, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886